CLINICAL TRIAL: NCT06345833
Title: Topical and Local TXA in Facelifts - A Randomized Controlled Double Blinded Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ENT-2024-32847
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Hemophilia; Hemorrhage; Facelift Surgery
MeSH Terms: conditions — Hemophilia A; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): 1% TXA mixed with standard local consisting 1/4% lidocaine with 1:100,000 epinephrine with saline as the control.
  Each face is treated as a split face and one half gets randomized to a TXA containing treatment group, so that each participant serves as his/her own control.
  Interventions: Drug: 1%Tranexamic acid with standard local
- Group 2 (Experimental): 3% TXA on TXA-soaked pledgets applied for 10 minutes with saline as the control
  Each face is treated as a split face and one half gets randomized to a TXA containing treatment group, so that each participant serves as his/her own control.
  Interventions: Drug: 3% TXA
- Group 3 (Experimental): 1% TXA with local plus 3% TXA-soaked pledgets with saline as the control
  Each face is treated as a split face and one half gets randomized to a TXA containing treatment group, so that each participant serves as his/her own control.
  Interventions: Drug: 1% TXA with local plus 3% TXA-soaked pledgets

INTERVENTIONS:
Drug: 1%Tranexamic acid with standard local — 1% TXA mixed with standard local consisting 1/4% lidocaine with 1:100,000 epinephrine with saline as the control.
  Arms: Group 1
Drug: 3% TXA — 3% TXA on TXA-soaked pledgets applied for 10 minutes with saline as the control.
  Arms: Group 2
Drug: 1% TXA with local plus 3% TXA-soaked pledgets — 1% TXA with local plus 3% TXA-soaked pledgets with saline as the control.
  Arms: Group 3

SUMMARY:
Tranexamic acid (TXA) is a fibrinolytic inhibitor which prevents prolonged bleeding by interfering with fibrin clot breakdown by competitively binding to lysine receptors on plasminogen; this prevents the conversion of plasminogen to plasmin. TXA will be applied to a randomly assigned side of the face during facelift surgery. The intervention groups will include 1% TXA mixed with standard local consisting 1/4% lidocaine with 1:100,000 epinephrine, 3% TXA on TXA-soaked pledgets applied for 10 minutes, and 1% TXA with local plus 3% TXA-soaked pledgets. Each treatment arm will be compared to saline in place of TXA on the contralateral side of the face.

Although TXA has been widely used in surgical fields for decades and is officially recommended by agencies such as ACOG for use during maternal hemorrhage, its current FDA approval only pertains to oral TXA for heavy menstrual bleeding and IV use for patients with hemophilia to prevent or reduce hemorrhage (cite). The main concern with intravenous TXA is the increased risk for the potential formation of blood clots, mainly in patients with clotting disorders, such as Facor V Leiden, and patients on estrogen containing medication. A recent systemic review with metanalysis by Wang et.al contained a total of 2150 patients receiving IV TXA while undergoing plastic surgery concluded that use of IV TXA does not lead to increased adverse events.[12] Given the low rate of adverse events while using TXA systemically, this protocol's application of TXA topically and/or locally negates the risk for any potential systemic adverse effects. No systemic adverse effects have been reported in studies examining local TXA in facial plastic surgery to date.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will consist of all regular clinic patients who elect and are deemed fit by the surgeon to undergo facelift surgery, including patients undergoing ancillary procedures
* age 18 and older
* English speaking.

Exclusion Criteria:

* younger than 18
* previously had an adverse reaction to tranexamic acid
* non-English speaking
* patients who elect not to participate or withdraw from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Blood loss | 2 weeks post-op
  measured through post-operative drain output, post-operative edema and ecchymosis.
  drain output is believed to be a more accurate representation of blood loss as it directly assesses the area in which TXA was applied as compared to intra-operative blood loss, which would be heavily influenced by bleeding from the skin incision.

SECONDARY OUTCOMES:
adverse effects of TXA rates | 2 weeks post-op
  in the form of flap epidermolysis, hair loss, or abnormal scar formation (e.g. hypertrophic scars) at the incision sites post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Jenna Van Beck, MD, Principal Investigator — University of Minnesota; Friederike Luetzenberg,, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States